CLINICAL TRIAL: NCT04195334
Title: Does Intramedullary Nail Diameter to Canal Ratio Predict the Incidence of Femoral Nonunion?
Brief Title: IMN Diameter to Femoral Canal Diameter and Union
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mina kamal, orthopedic resident doctor mina kamal kamel, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMN diameter and union
Record Dates: First submitted 2019-11-28; First posted 2019-12-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2019-12

CONDITIONS: Femoral Shaft Fracture
Keywords: intramedullary nail

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMN and union (Experimental): putting an intramedullary nail in femoral shaft fractures and finding a relation between the nail diameter to femoral canal diameter and how this will affect healing or predict union
  Interventions: Device: internal fixation by IMN

INTERVENTIONS:
Device: internal fixation by IMN — using retrograde or antegrade IMN for femooral fractures fixation using a fit nail to the femoral intramedullary canaland follow up for union

SUMMARY:
To Detect the Relation Between the Intramedullary Nail Diameter to Canal Ratio and the Incidence of Non-union

DETAILED DESCRIPTION:
Femoral intramedullary nail fixation is currently considered the ''gold standard'' for treatment of femoral shaft fractures in adult population. Clinical outcomes after operative treatment of proximal femur fracture have been shown to be dependent on achieving optimal mechanical alignment and union. Patient independent risk factors associated with nonunion after intramedullary fixation includes: open fracture, undreamed intramedullary nailing, fracture comminution, non-isthmal and particularly infra-isthma fracture location and infection. Patient dependent risk factors include smoking, diabetes, nonsteroidal anti-inflammatory medications, closed head injury and delayed weight. Unreamed nailing allows for better maintenance of the endosteal circulation at the expense of smaller diameter implants; in contrast, reamed applications permit a larger diameter nail, resulting in stronger fixation constructs and earlier fracture union. After reaming, a larger diameter intramedullary nail is placed. When initially reported, this treatment resulted in high success rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age (20_60) years old
2. Closed fracture and open grade one
3. Midshaft fractures type3\2 according to the OA classification
4. pattern of the fracture (simple transverse,oblique ,spiral)
5. Retrograde and Antigrade nail

Exclusion Criteria:

1. Open fractures grade two and three.
2. patient with comorbidities eg(DM.HTN…)
3. severe osteoporosis with wide medulla .
4. patient on regular steroid therapy.
5. patient refused to be enrolled in the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The ratio between IMN and femoral canal diameter and incidence of union objectively | 6 months
  We will measure union objectively using x ray (union in 3 or more cortices)
measurement of union clinically | 6 months
  we will measure the union clinically using visual analog score after 6 weeks.( Change From Baseline in Pain Scores on the Visual Analog Scale at 6 Weeks).
  then we will test if there is a relation between union and the ratio between femoral canal and IMN diameter.

CONTACTS AND LOCATIONS:
Overall Officials: ALY MOHAMADEEN, MD, Study Chair — Assiut University; mahmoud badran, MD, Study Director — Assiut University

REFERENCES:
- [Background] Millar MJ, Wilkinson A, Navarre P, Steiner J, Vohora A, Hardidge A, Edwards E. Nail Fit: Does Nail Diameter to Canal Ratio Predict the Need for Exchange Nailing in the Setting of Aseptic, Hypertrophic Femoral Nonunions? J Orthop Trauma. 2018 May;32(5):245-250. doi: 10.1097/BOT.0000000000001110. PMID 29401087
- [Background] Shroeder JE, Mosheiff R, Khoury A, Liebergall M, Weil YA. The outcome of closed, intramedullary exchange nailing with reamed insertion in the treatment of femoral shaft nonunions. J Orthop Trauma. 2009 Oct;23(9):653-7. doi: 10.1097/BOT.0b013e3181a2a337. PMID 19897987
- [Background] Rudloff MI, Smith WR. Intramedullary nailing of the femur: current concepts concerning reaming. J Orthop Trauma. 2009 May-Jun;23(5 Suppl):S12-7. doi: 10.1097/BOT.0b013e31819f258a. PMID 19390369
- [Background] Collinge CA, Hymes R, Archdeacon M, Streubel P, Obremskey W, Weber T, Watson JT, Lowenberg D; Members of the Proximal Femur Working Group of the Southeast Trauma Consortium. Unstable Proximal Femur Fractures Treated With Proximal Femoral Locking Plates: A Retrospective, Multicenter Study of 111 Cases. J Orthop Trauma. 2016 Sep;30(9):489-95. doi: 10.1097/BOT.0000000000000602. PMID 27144821